CLINICAL TRIAL: NCT06987682
Title: Stimulating Postural Control to Augment Rehabilitation After Cerebral Stroke (SPARC): a Pilot Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 24-5792
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: functional electrical stimulation; transcutaneous spinal cord stimulation; postural control
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance training + transcutaneous spinal stimulation (Experimental)
  Interventions: Other: Balance training
- Balance training + sham transcutaneous spinal stimulation (Sham Comparator)
  Interventions: Other: Balance training

INTERVENTIONS:
Other: Balance training — Participants will don a safety harness that is secured to an overhead track. Each balance training session will involve 60 minutes of reactive balance training (RBT). For both intervention arms, trancutaneous spinal stimulation will be set up, including placing electrodes and setting stimulation amplitudes.

SUMMARY:
People living with stroke have a high risk of falling and this risk increases as mobility improves over the first year post-stroke. Despite the high number of falls, there is a lack of interventions to prevent falls after stroke. One possible solution is to alter nerve activity through delivery of a stimulus, such as electrical stimulation. The purpose of this study is to test the study plan and to find out whether enough participants will join a larger study and accept the study procedures of combining electrical stimulation with balance training.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or greater
* Diagnosed with a middle cerebral artery stroke >1 year ago
* Community-dwelling (i.e. not living in long-term care or other inpatient setting)
* Able to stand independently for 60 seconds
* Able to understand spoken English

Exclusion Criteria:

* Any condition other than stroke that significantly affects their postural control (e.g. vestibular disorder, vision loss)
* A prior lower extremity fragility fracture
* A planned injection of botulinum toxin to the legs during the intervention period
* Peripheral nerve damage in the legs
* Contraindications for electrical stimulation (i.e. implanted electronic device, active cancer or radiation in past six months, uncontrolled epilepsy, skin rash/wound at an electrode site, pregnancy, active deep vein thrombosis)
* Contraindications for TMS (i.e. seizures, metal in the head)
* Previous participation in tSCS within the past 2 years (May affect blinding integrity. Likely uncommon; FES is rarely used in Canada post-stroke.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mini-Balance Evaluation Systems Test | From enrollment to the 12-week post-intervention follow-up
Activities-specific Balance Confidence Scale | From enrollment to the 12-week post-intervention follow-up

SECONDARY OUTCOMES:
Gait and standing spatiotemporal data | From enrollment to the 12-week post-intervention follow-up
  Collected using the Zeno Walkway Gait Analysis System
Corticospinal excitability of the affected soleus and tibialis anterior | From enrollment to the 12-week post-intervention follow-up
  TMS will be delivered using a magnetic stimulator with a double-cone coil

CONTACTS AND LOCATIONS:
Locations (1):
- KITE Research Institute, Toronto Rehabilitation Institute - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided